CLINICAL TRIAL: NCT00565630
Title: Pilot Study on Bioavailability of Vigamox Administered as Drops vs. as Spray
Brief Title: Using Device Delivering Ophthalmic Solution in a Spray Form Instead of Eye Drops
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Replaced with ongoing study
Sponsor: Advanced Ophthalmic Pharma (Industry)
Responsible Party: Principle Investigator: Dr. Adi Michaeli, Dept. of Ophthalmology, TAMC, Tel Aviv, Israel
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Drops vs. spray administration; TAMC 06-306
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2007-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Vigamox via the experiemntal device
  Interventions: Device: Vigamox delivered via the device in spray form
- 2 (Active Comparator): Vigamox drops from the commercially available bottles
  Interventions: Device: Vigamox delivered via the device in spray form

INTERVENTIONS:
Device: Vigamox delivered via the device in spray form — Vigamox delivered 4 times, 1 hour prior to cataract surgery

SUMMARY:
The purpose of the study is to confirm that Vigamox reaches similar aqueous concentration when administered as the commercially available eye drops or as a spray delivered from a proprietary device.

DETAILED DESCRIPTION:
Patients scheduled for elective cataract surgery, will be randomly allocated to receive Vigamox 4 times , 1 hour prior to surgery, either via the experimental device in a spray form, or via the regular, commercially available bottle.

Aqueous sample will be collected and submitted to a masked laboratory for measuring Vigamox concentration.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cataract surgery

Exclusion Criteria:

* Known allergy to quinolone compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-01; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Aqeous concentration of Vigamox | one month

CONTACTS AND LOCATIONS:
Overall Officials: Adi Michaeli, MD, Principal Investigator — Dept of Ophthalmology, TAMC, Tel Aviv, Israel